CLINICAL TRIAL: NCT01781351
Title: Neuromuscular Control of the Ankle With External Support
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Dr. med. Benita Kuni, MD, Dr. med B. Kuni, University Hospital Heidelberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 407- 05_121126
Record Dates: First submitted 2013-01-15; First posted 2013-02-01 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Chronic Ankle Instability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- taping the ankle (Experimental)
  Interventions: Other: Taping the ankle

INTERVENTIONS:
Other: Taping the ankle

SUMMARY:
Untreated ankle sprains often remain symptomatic and may end in chronic instability. The aim of our study is to quantify the stabilizing effect of different devices. Through the combined use of the 3D motion analysis and the surface electromyography, the influence of the devices with respect to a mechanical effect and to an influence on the neuromuscular control are examined. The tests will simulate situations with a higher risk of injury. In the experimental set-up, an element of surprise will be integrated in order to analyze any muscular compensation mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* chronic ankle instability
* "giving way"
* repeated ankle sprains

Exclusion Criteria:

* other injuries of the lower extremities
* surgery on the lower extremities

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Change in elektromyographic signal in peroneus longus muscle (surface EMG) | baseline (=before) and immediately after applying the device

CONTACTS AND LOCATIONS:
Overall Officials: Benita Kuni, Dr. med., M.D., Principal Investigator — Dep. of Orthopedics, Trauma Surgery and Spinal Cord Injury
Locations (1):
- Department of Orthopedics, Trauma Surgery and Spinal Cord Injury, Heidelberg University Hospital, Heidelberg, Germany